CLINICAL TRIAL: NCT01365741
Title: Time to Thrombocytic Inhibition After Supine and Upright Ingestion of Efient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jacob Antonsen, Medical Doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TTISUE
Record Dates: First submitted 2010-12-21; First posted 2011-06-03 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Heart Disease; Ischemic Heart Disease; ST-elevation Myocardial Infarction
Keywords: PCI; STEMI; Interventions; Heart disease; Thrombocytic inhibition; Cross-over study; Percutaneous coronary intervention
MeSH Terms: conditions — Heart Diseases; Myocardial Ischemia; ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard administration of Efient (No Intervention): The test person will ingest Efient in supine position, and remain supine during 2 hours, mimicing the way Efient is used for pre-PCI treatment today
- Upright administration of Efient (Active Comparator): The test person will ingest Efient in an upright position, and remain supine during 2 hours.
  Interventions: Other: Upright position

INTERVENTIONS:
Other: Upright position — The test person will ingest Efient in an upright position and remain upright for 2 minutes. After 2 minutes, the test person will lie down, and remain supine for 2 hours, the same way as the person did in the control arm
  Other Names: Efient; Prasugrel; PCI
  Arms: Upright administration of Efient

SUMMARY:
The purpose of the study is to clarify wether body posture during ingestion of 60mg Efient, a thrombocytic inhibitor, has influence on the time to thrombocytic inhibition.

The study aims to mimic the treatment Danish patients receive when admitted to the hospital with a ST-elevation myocardial infarction since these patients are refereed to acute Percutaneous Coronary Intervention (PCI) necessitating fast and efficient thrombocytic inhibition.

Current guidelines recommend the administration of Efient right before the PCI procedure, while the patient is lying down, either in the ambulance or in the operating room. We, the investigators, believe that this is suboptimal for the patient, since any sort of prolonged inhibition time will possibly worsen the patients prognosis and make the patient more prone to later clotting issues.

Our hypothesis is that by making the patients ingest the tablets in a 90 degrees upright position and making them sit up for 2 minutes after ingestion, the effect of the pills will commence faster than if taken in a supine position. This will possibly lead to faster inhibition of the thrombocytes, which we believe will lead to a lower incidence of clotting issues during and after the procedure.

DETAILED DESCRIPTION:
The study will be divided into two sessions: first session will be the control arm- ingestion of Efient in supine position.

14 days later, the same test-persons will be doing the intervention- ingestion of Efient sitting upright for 2 minutes. Besides this, the second session will be exactly the same as the control arm.

ELIGIBILITY:
Inclusion Criteria:

* 20-30 years of age
* Healthy
* Male
* Ability to give informed consent
* Non-Smoker

Exclusion Criteria:

* Known with reflux or dysphagia
* Ingestion of medicine, beside Paracetamol <14 prior to the trial
* Hematological diseases
* Diabetes
* Known kidney disease
* Known liver disease
* Recent trauma
* Scheduled operation within 7 days after the trial
* Former apoplexia
* Known gastro-intestinal disease
* Weight <60 kg

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Inhibition of ADP-receptors on thrombocytes | Blood will be drawn from the test person at 0, 20, 40, 60, 80, 100minutes post ingestion.
  The primary outcome will be the difference between the time to sufficient/maximal inhibition of the ADP-receptors on the test-persons thrombocytes compared between supine and upright ingestion of Efient.
  Inhibition will be verified bedside by VerifyNow analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Antonsen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antonsen J, Bundgaard N, Holmvang L, Engstrom T, Iversen K. Posture changes platelet inhibition time after ingestion of prasugrel. Dan Med J. 2018 Oct;65(10):A5504. PMID 30269747
- See also: Related Info — http://ugeskriftet.dk/dmj/posture-changes-platelet-inhibition-time-after-ingestion-prasugrel